CLINICAL TRIAL: NCT06798701
Title: Symptom Management in the Bone Marrow Transplant Patient Population Using Virtual Reality
Brief Title: Virtual Reality for Symptom Management in Patients Undergoing Hematopoietic Stem Cell Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: I-4062924; NCI-2024-10766 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I-4062924 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2025-01-22; First posted 2025-01-29 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm I (VR use) (Experimental): Patients use the VR device to participate in applications related to relaxation such as mediation, art and nature, for up to 15 minutes, daily, while inpatient for standard of care HSCT.
  Interventions: Other: Interview; Other: Survey Administration; Procedure: Virtual Reality
- Arm II (Standard care) (Active Comparator): Patients undergo standard care for the HSCT.
  Interventions: Other: Best Practice; Other: Survey Administration

INTERVENTIONS:
Other: Best Practice — Undergo standard care
  Other Names: standard of care; standard therapy
  Arms: Arm II (Standard care)
Other: Interview — Ancillary studies
  Arms: Arm I (VR use)
Other: Survey Administration — Ancillary studies
Procedure: Virtual Reality — Use VR device
  Other Names: VR
  Arms: Arm I (VR use)

SUMMARY:
This clinical trial compares the use of virtual reality to standard care for improving symptom management in patients undergoing hematopoietic stem cell transplantation (HSCT). Significant symptoms experienced by hospitalized HSCT patients include, but are not limited to, depression, tiredness, anxiety, drowsiness, lack of appetite, pain, and overall decreased quality of life and well-being. Virtual reality (VR) as an intervention can provide these patients with a much-needed escape from their reality and has proven results in clinical settings as a distraction therapy. VR technology targets the patient's auditory, visual, and physical contact/touch senses, and has been evidenced to improve depression, fatigue, anxiety, appetite, and pain. Virtual reality may improve symptom management in patients undergoing HSCT.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the efficacy of VR for symptom management in the admitted HSCT patient population.

SECONDARY OBJECTIVE:

I. To examine the use of supportive medications for symptom management after HSCT while using VR.

EXPLORATORY OBJECTIVE:

I. To evaluate any limitations or barriers of the use of VR in the inpatient setting throughout the study.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients use the VR device to participate in applications related to relaxation such as mediation, art and nature, for up to 15 minutes, daily, while inpatient for standard of care HSCT.

ARM II: Patients undergo standard care for the HSCT.

After completion of study intervention, patients are followed up after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old) admitted to Roswell Park on 5 North for planned hematopoietic stem cell transplantation (HSCT)
* Must be alert and oriented (Glascow Coma Scale of 15, Nursing Universal Flowsheet) and able to consent to participate in the study
* Expected to be admitted to Roswell Park inpatient unit for ≥ 1 week
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant patients
* Incarcerated patients
* Patients who are unwilling or unable to follow protocol requirements
* Individuals that are prone to motion sickness, nausea, dizziness, history of seizure, potential for seizure, history of delirium, at risk for confusion, etc
* Participants with audio and/or visual impairments that would preclude them from using a VR device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2026-03-14 (Estimated); Study Completion 2026-03-14 (Estimated)

PRIMARY OUTCOMES:
Difference in the trajectories of the mean Edmonston Symptom Assessment System Revised (ESAS-r) composite scores | Length of hospital stay up to 6 months
  Firstly, the pattern of ESAS-r scores over time will be graphically examined. To account for the within-individual correlations, a generalized linear mixed model with appropriate link function will be applied. The time is measured by the number of days after treatment start and will be considered as a continuous variable. The effect of interest is the time by group interaction. Significant interaction implies different trajectories of ESAS-r composite scores over time. If the nonlinear patterns were observed, appropriate transformation or analyses focusing on the linear region will be considered. All tests will be two sided at a significant level of 0.05. Scores of individual items will be compared using the same approach. False discovery rate will be controlled using Benjamini-Hochberg procedure. As complementary analyses, models with only surveys before or after the virtual reality will also be examined.

SECONDARY OUTCOMES:
Counts of supportive medication administration | Length of hospital stay up to 6 months
  Will be compared between two arms using generalized linear mixed models with appropriate link functions. The types of medications will be summarized by counts and percentages for each arm. Pre-intervention counts will be compared to during-intervention counts. The types of supportive medications will also be examined (i.e. anxiolytic, antidepressant, analgesic or antiemetics). Medications include (but are not limited to) the following: hydromorphone, acetaminophen, lorazepam, ondansetron, prochlorperazine, trazodone, and tramadol.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Huizinga, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States